CLINICAL TRIAL: NCT00858650
Title: Registry of Hypogonadism in Men
Acronym: RHyMe
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: Bayer (Industry); Besins Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: RHyMe
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-04

CONDITIONS: Male Hypogonadism; Androgen Deficiency; Testosterone Deficiency
Keywords: registry; natural history
MeSH Terms: conditions — Eunuchism | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard of Care: Hypogonadal males treated by standard of care, with or without testosterone replacement therapy
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Standard of care may or may not include use of testosterone replacement therapy

SUMMARY:
The primary objective of the Registry of HYpogonadism in MEn (RHYME) is to establish and maintain a large, multi-national prospective registry of male patients who have been diagnosed with male hypogonadism (HG), also known as androgen deficiency or testosterone deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18 years and older.
2. Diagnosis of hypogonadism including Klinefelter's or late onset HG. Patients may have been diagnosed at any point in their lives. Documentation of the diagnosis of HG (including symptomatology and laboratory values including testosterone levels confirmed on two separate occasions) is required.
3. Written informed consent.

Exclusion Criteria:

1. Any previous treatment with testosterone therapy.
2. History of breast cancer, prostate cancer, or high-grade prostatic intraepithelial neoplasia.
3. Prior radical prostatectomy.
4. Life expectancy shorter than 24 months as judged by the Clinical Site investigator.
5. Current major psychiatric disorders or drug or alcohol abuse, which will likely affect participation or compliance in the Registry, in the opinion of the Clinical Site Investigator.
6. Gender dysphoria or sexual reassignment (e.g., transexualism).
7. Patients actively enrolled in any interventional clinical trial.
8. Planned relocation outside Clinical Site region within 24 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypogonadal men
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Prostate Cancer | 2-years

SECONDARY OUTCOMES:
PSA, IPSS, and Other Urologic Outcomes | 3-years
Sexual Function and Hypogonadism Symptoms | 3-years
Physical Health and Cardiovascular Outcome Measures | 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Rosen, PhD, Principal Investigator — New England Research Institutes, Inc
Locations (25):
- Germany (4):
  - University Hospital Halle - Center for Reproductive Medicine and Andrology, Halle
  - Institute of Urology and Andrology, Segeberger Kliniken, Hamburg
  - Private Practice of Andrology & Urology, Hamburg
  - Klinik fur Innere Medizin,, Herne
- Italy (5):
  - Ospedali Riuniti, Ancona
  - Unità di Andrologia DFC AziendaOspedalieraUniversitariaCareggi, Florence
  - Hesperia Hospital, Modena
  - University of Parma, Parma
  - University of Rome - Sapienza, Rome
- Netherlands (4):
  - Amstelland Hospital, Amstelveen
  - VU medical centre, department of Urology, Amsterdam
  - Andros Men's Health Institutes, Arnhem
  - Erasmus Medical Center - Urology, Rotterdam
- Spain (5):
  - Fundacio Puigvert, Barcelona
  - Hospital Universitario doce de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro- Majadahonda, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen del Rocio, Seville
- Sweden (2):
  - Urohälsan i Skövde: Gotenborg University, Gotenborg
  - Karolinska University Hospital - Centre for Andrology and Sexual Medicine, Stockholm
- United Kingdom (5):
  - Barnsley Hospital, Barnsley
  - Royal Free Hospital, Hampstead
  - Holly Cottage Clinic, Lichfield
  - Manchester Royal Infirmary, Manchester
  - Royal Victoria Infirmary, Newcastle